CLINICAL TRIAL: NCT03492268
Title: Safety and Efficacy Evaluation of Autologous BCMA-CART for Treating Relapsed or Refractory Multiple Myeloma
Brief Title: Safety and Efficacy Evaluation of BCMA-CART for Treating Multiple Myeloma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to CART processing facility construction
Sponsor: Bioray Laboratories (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-CART-00CH3(1)
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Patients undergo leukapheresis to separate their lymphocytes, from which CART cells are produced. Patients will receive a conditioning therapy with cyclophosphamide and fludarabine before CART therapy. BCMA-CART cells will be injected intravenously (IV) into patients on day 0.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA-CART (Experimental): Autologous T cells transduced to express anti-BCMA chimeric antigen receptor (CAR)
  Interventions: Biological: BCMA-CART

INTERVENTIONS:
Biological: BCMA-CART — After a conditioning therapy, each patient will receive a treatment of BCMA-CART originated from their own peripheral blood mononuclear cells

SUMMARY:
This trial aims to evaluate the safety and efficacy of BCMA-CART in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
BCMA(B-Cell maturation antigen) is a tumor antigen of multiple myeloma . Using a genetic engineering strategy to assemble an anti-BCMA CAR(chimeric antigen receptor) in autologous T cells will help these CART cells to recognize and kill BCMA-expressing MM tumor cells. This trial aims to evaluate the safety and anti-tumor efficacy of autologous BCMA-CART in treating relapsed or treatment refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Have the capacity to give informed consent;
* Confirmed diagnosis of active MM as defined by NCCN and IMWG criteria;
* Have a diagnosis of BCMA+ multiple myeloma (MM), (≥ 5% BCMA+ in CD138+ plasma cells by flow cytometry obtained within 45 days of study enrollment);
* Refractory and relapsed MM patients after > 2 cycles of induction therapy,or,have relapsed or treatment refractory disease following autologous stem cell transplant (ASCT);
* ECOG score=0-2.

Exclusion Criteria:

* Pregnant or nursing women; Women of reproductive potential must have a negative serum pregnancy test performed within 48 hours of starting conditioning chemotherapy;
* Active infection, HIV infection, syphilis serology reaction positive;
* Active hepatitis B, hepatitis C at the time of screening;
* Significant hepatic dysfunction as following, SGOT(serum glutamic-oxaloacetic transaminase)> 5 x upper limit of normal; bilirubin > 3.0 mg/dL;
* Lymphotoxic chemotherapeutic agents within 2 weeks of leukapheresis serious mental disorder;
* With severe cardiac, liver, renal insufficiency, diabetes and other diseases;
* Participate in other clinical research in the past three months; previously treatment with any gene therapy products;
* Contraindication to cyclophosphamide or fludarabine chemotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 90 days after T cell infusion
  Proportion of patients in whom a response among complete response or partial response, as defined by International Myeloma Working group(IMWG) response criteria , will be observed.

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events as a Measure of Safety | Baseline up to 35 days
  Adverse events assessed according to NCI-CTCAE v4.03 criteria
Duration of persistence of BCMA-CART | Baseline up to 1 year
  BCMA-CART duration be assessed by FACS or QPCR

CONTACTS AND LOCATIONS:
Overall Officials: Yunxiao Xu, MD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- Shanghai Bioray Laboratories INC., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No